CLINICAL TRIAL: NCT01974557
Title: The Effect of Age on the Hemodynamic Response During Rest and Exercise in Healthy Humans
Acronym: HemReX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finn Gustafsson (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2-2013-072
Record Dates: First submitted 2013-10-22; First posted 2013-11-01 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Hemodynamics
Keywords: Cardiac physiology; ageing; gender differences; diastole; fluid challenge
MeSH Terms: conditions — Heart Murmurs | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Exercise

SUMMARY:
Primary: To observe how hemodynamic parameters are affected by age during rest and exercise in healthy humans. Furthermore, how an acute fluid challenge changes hemodynamic parameters.

Secondary: To thoroughly examine this population with regard to cardiac performance and function, anthropometrics, metabolic status, exercise capability, constitution, pulmonary status, and humoral markers of organ functions. This population will serve as a healthy control group, to which different populations can be compared, hence the need for a comprehensive characterization.

Hypotheses:

Diastolic function and parameters associated with diastolic function gradually deteriorate with increasing age. The gradual deterioration is unmasked at an earlier age during exercise and fluid challenge, compared to measurements made at rest.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* No acute or chronic diseases that can influence hemodynamics
* Pause in medication with effect on hemodynamics 24h before experimental day
* Echocardiography, with no structural abnormalities with an impact on hemodynamics.
* ECG without any pathological findings, including arrhythmia
* Normal red and white blood count, normal renal, liver, thyroid, immune, and hematological function as well as normal electrolytes, HbA1c and natriuretic peptides
* Ability to perform graded bicycle exercise testing
* BMI in the range of 20-30 kg/m2
* Height within population mean ±2 standard deviations
* VO2-max within population mean ±2 standard deviations (age corrected)
* Acceptable sonographic conditions
* Informed consent

Exclusion Criteria:

* History of heart failure (verified or suspected), or heart failure verified by pathological left and right systolic and diastolic measurements of the heart
* Hypotension (systolic blood pressure < 100 mmHg)
* Inability to participate
* Pregnant women
* Diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Composite of hemodynamic parameters | minutes
  Invasive measurements using Swan-Ganz catheters and echocardiography will provide the data needed.

SECONDARY OUTCOMES:
Composite of humoral markers | up to 1 hour
  Blood samples will be analysed with regard to humoral peptides and hormones that may affect hemodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, M.D. Msc, Principal Investigator — Chief Physician
Locations (1):
- Dept. of Cardiology, Rigshospitalet, University Hospital of Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen MJ, Wolsk E, Bakkestrom R, Christensen N, Carter-Storch R, Omar M, Dahl JS, Frederiksen PH, Borlaug B, Gustafsson F, Hassager C, Moller JE. Pressure-flow responses to exercise in aortic stenosis, mitral regurgitation and diastolic dysfunction. Heart. 2022 Nov 10;108(23):1895-1903. doi: 10.1136/heartjnl-2022-321204. PMID 36356959
- [Derived] Andersen MJ, Wolsk E, Bakkestrom R, Thomsen JH, Balling L, Dahl JS, Gustafsson F, Moller JE, Hassager C. Hemodynamic Response to Rapid Saline Infusion Compared with Exercise in Healthy Participants Aged 20-80 Years. J Card Fail. 2019 Nov;25(11):902-910. doi: 10.1016/j.cardfail.2019.06.004. Epub 2019 Jun 17. PMID 31220623